CLINICAL TRIAL: NCT05906810
Title: Impact of Non-surgical Periodontal Therapy in the Improvement of Early Endothelial Dysfunction in Subjects With Peri-implantitis and Peri-implant Mucositis: a Randomized-controlled Clinical Trial.
Brief Title: Impact of Non-surgical Periodontal Therapy in the Improvement of Early Endothelial Dysfunction in Subjects With Peri-implantitis and Peri-implant Mucositis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 121-23
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Atherosclerosis; Endothelial Dysfunction; Peri-Implantitis; Peri-implant Mucositis
MeSH Terms: conditions — Atherosclerosis; Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: The main objective of this study is to evaluate the efficacy of periodontal treatment on the improvement in cardiovascular parameters.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Peri-implantitis (Experimental): Subjects diagnosed with peri-implantitis according to the most recent international guidelines and without cardiovascular diseases.
  Interventions: Procedure: Non-surgical periodontal treatment
- Peri-implant mucositis (Active Comparator): Subjects diagnosed with peri-implant mucositis according to the most recent international guidelines and without cardiovascular diseases.
  Interventions: Procedure: Non-surgical periodontal treatment
- Healthy (No Intervention): Subjects without periodontitis and with good gingival health.

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Subgingival biofilm ultrasonic debridement
  Arms: Peri-implant mucositis; Peri-implantitis

SUMMARY:
A double-blind randomized-controlled clinical trial is conducted in order to evaluate the impact of non-surgical periodontal treatment on endothelial dysfunction parameters in subjects with peri-implantitis/peri-implant mucositis and without any cardiovascular disease.

DETAILED DESCRIPTION:
A double-blind randomized-controlled clinical trial is conducted in order to evaluate the impact of non-surgical periodontal treatment on endothelial dysfunction parameters in subjects with peri-implantitis/peri-implant mucositis and without any cardiovascular disease.

90 patients: 30 with peri-implantitis, 30 with peri-implant mucositis and 30 healthy controls and without periodontitis history.

All the patients are assessed for clinical, periodontal, blood and non-invasive ultrasound cardiovascular parameters. Measurements are taken before and after initial periodontal treatment in the peri-implantitis/peri-implant mucositis subjects.

ELIGIBILITY:
PERI-IMPLANTITIS GROUP

Inclusion Criteria:

• Clinically diagnosed with peri-implantitis according to the EFP/AAP 2017 criteria.

Exclusion Criteria:

* Periodontal treatment, implant surgery, antibiotics, NSAIDs, immunosuppressants during the last 6 months.
* Pregnancy.
* Cardiovascular Diseases.

PERI-IMPLANT MUCOSITIS GROUP

Inclusion Criteria:

• Clinically diagnosed with peri-implant mucositis according to the EFP/AAP 2017 criteria.

Exclusion Criteria:

* Periodontal treatment, implant surgery, antibiotics, NSAIDs, immunosuppressants during the last 6 months.
* Pregnancy.
* Cardiovascular Diseases.

HEALTHY GROUP

Inclusion Criteria:

• Clinically diagnosed with healthy periodontum withouth periodontitis history according to the EFP/AAP 2017 criteria.

Exclusion Criteria:

* Scaling, antibiotics, NSAIDs, immunosuppressants during the last 6 months.
* Pregnancy.
* Cardiovascular Diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Velocity carotid-femoral (PWV-CF) | 8 weeks
  The speed of pulse wave propagation between carotid-femoral sites
Pulse Wave Velocity carotid-femoral (PWV-CR) | 8 weeks
  The speed of pulse wave propagation between carotid-radial sites
Carotid Intima-Media Thickness (CIMT) | 8 weeks
  The thickness of the carotid intima and media
Distensibility Coefficient (DC) | 8 weeks
  The relative change in luminal area during systole for a given pressure change (pulsed pressure), will be calculated assuming the lumen to be circular.
Advanced Glycation End products (AGEs) | 8 weeks
  A group of endogenous heterogeneous compounds that are constantly formed under physiological conditions with prooxidant and cytotoxic properties. Measurements are performed by fluorescence spectroscopy technique.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: No